CLINICAL TRIAL: NCT02869399
Title: A Randomized Phase II Study for Tertiary Prevention of Squamocellular Cancer of Head and Neck (SCCHN) With a Dietary Intervention
Brief Title: Tertiary Prevention of Head and Neck Cancer With a Dietary Intervention
Acronym: DietINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INT 18/15
Record Dates: First submitted 2016-08-11; First posted 2016-08-17 (Estimated); Last update posted 2023-03-13 (Actual); Status verified 2022-04

CONDITIONS: Cancer of Head and Neck
Keywords: head and neck cancer, nutritional intervention
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental arm (Experimental): The experimental arm is based on a dietary intervention in addition to standard recommendations.The diet will be based on the AICR/WCRF recommendations for cancer prevention and for the prevention of recurrences. The intervention strategy will focus on reducing inflammation and reducing glycaemia and insulinaemia while promoting nutrient-rich diet. Patients will be taught how to prepare traditional Mediterranean meals (healthy, satiating, palatable and easy to prepare).
  Interventions: Dietary Supplement: dietary intervention in addition to standard recommendations
- Control arm (No Intervention): Patients in the control arm will not receive specific suggestions concerning diet, but standard healthy lifestyle recommendations will be given. The recommendations, including nutritional consultation if needed by standard practice of care, will be reinforced at each clinical visit and through a leaflet according to primary cancer prevention nutritional guidelines. Patients in the control group will not receive any of the recipes or educational materials given to the intervention group and they will not have kitchen classes.

INTERVENTIONS:
Dietary Supplement: dietary intervention in addition to standard recommendations — The diet of the intervention group will be based on the AICR/WCRF recommendations for cancer prevention and for the prevention of recurrences (www.dietandcancerreport.org):
  * avoid or limit alcoholic drinks (2 drinks men, 1 drink women)
  * increase consumption of a variety of non-starchy vegetables, fruits (at least 400g per day) and dietary fibers (at least 25g per day)
  * eat mostly food of plant origin
  * eat lean meat, limit intake of red meat and avoid processed meat
  * increase consumption of anti-inflammatory foods, such as fish and whole grain cereals, f.e. brown rice and barley creams
  * avoid high glycaemic and high insulinemic foods, such as refined flours, white breads, and pastries
  Arms: Experimental arm

SUMMARY:
This is an open-label randomized phase II multicenter trial. An estimated 350 patients deemed to be in complete remission at month 3 after curative treatment are considered for this trial. Two arms of intervention are foreseen: the experimental arm (arm A) based on dietary intervention in addition to standard recommendations and a control arm (arm B) including only standard recommendations. The intervention strategy is based on the AICR/WCRF recommendations for cancer and recurrences prevention and it is focused on decreasing inflammation, glycaemia and insulinaemia while promoting nutrient-rich diet. The reduction in the incidence of tumor recurrence will be analyzed comparing EFS curves between the two arms with the non-parametric Kaplan-Meier method. Secondary analyses will describe the time trend in the prevalence of side effects and quality of life, as assessed by the EORTC QLQ-H&N35 questionnaire. Translational analysis (cytokine, salivary and plasmatic miRNA) will be performed. The trial is coordinated by Istituto Nazionale Tumori, Milan and conducted in 6 European countries.

DETAILED DESCRIPTION:
Patients deemed to be in complete remission at month 3 (+/- 1 month) after curative treatment will be considered for this trial.

At each follow up visit the patients will state all the changes and new symptoms they experienced and they will receive both physical and fiberoptic endoscopic head and neck examination. Locoregional imaging should preferentially be performed within 6 months after treatment end and then will be recommended only on the occurrence of new signs or symptoms. Late adverse events of the treatment will be evaluated at each visit according to Common Toxicity Criteria of Adverse Events (CTCAE version 4.0). Quality of life questionnaire (EORTC QLQ HN35) and VSAQ questionnaire will be administered to patients every other visit. Laboratory tests including a complete blood count, renal, hepatic and thyroid function will be performed once a year. The analysis of blood biomarkers of compliance and efficacy will be conducted at baseline, 3, 6, 12, 18 and 24 months after randomization.

The proposed study foresees two arms of intervention: the experimental arm based on dietary intervention in addition to standard recommendations and a control arm which includes only standard recommendations.

The intervention strategy will focus on reducing inflammation and reducing glycaemia and insulinaemia while promoting nutrient-rich diet.

Patients will be taught how to prepare traditional Mediterranean meals (healthy, satiating, palatable and easy to prepare).

Patients in the control arm will not receive specific suggestions concerning diet, but standard healthy lifestyle recommendations will be given. The recommendations, including nutritional consultation if needed by standard practice of care, will be reinforced at each clinical visit and through a leaflet according to primary cancer prevention nutritional guidelines. Patients in the control group are encouraged to follow the WCRF/AICR recommendations but they will not receive any of the recipes or educational materials given to the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* High-risk effectively cured stage III and IV HNSCC
* Oropharyngeal cancer will be enrolled only if with a smoking history of more than 10 pack/years
* Able to swallow at least a soft pureed diet
* Male or female > 18 years
* Signed written informed consent

Exclusion Criteria:

* Serious or uncontrolled co-existent non-malignant disease, including active and uncontrolled infection
* Non parotid-sparing RT
* Severely malnourished patients (patients with a weight loss greater that 5% in the last month before enrollment and with a BMI < 20)
* Diabetic patients in pharmacological treatment
* Participation in clinical trials with other experimental agents within 30 days of study entry or concomitant treatment with other experimental drug
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study
* Other significant disease that in the investigator's opinion would exclude the subject from the trial
* Patients unable to comply with the protocol, in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2015-11; Primary Completion 2018-11 (Actual); Study Completion 2023-02 (Actual)

PRIMARY OUTCOMES:
Reduction in the incidence of tumor recurrence and second primaries | 36 months
  Reduction in the incidence of tumor recurrence and second primaries will be assessed. When a clinical or radiological evidence of recurrence exists, all the efforts should be made in order to perform a histological confirmation. It is possible that a certain amount of recurrences will not be cyto/histologically confirmed due to tumor location not making the sampling feasible. It will be accepted a maximum percentage of 10% of such cases, if in presence of at least 2 different concordant radiological imaging.
Identification of saliva and plasma miRNAs and evaluation of their change in the 2 arms of treatment | 36 months
  The project involves the monitoring of miRNAs during the dietary intervention to ascertain the effectiveness of the treatment and the relationship with clinical outcome
Change in inflammatory cytokine profile during the course of dietary intervention | 36 months
  The change in inflammatory cytokine profile during the course of dietary intervention and the comparison with control arm will be evaluated

SECONDARY OUTCOMES:
Reduction of treatment related side effects | 36 months
  Reduction of treatment related side effects (e.g. xerostomia, fatigue, mucositis), assessed according to CTCAE v 4.0 (physician assessed symptoms) will be evaluated during study course.
EORTC HN35 quality of life scales | 36 months
  The improvement of Quality of Life assessed according to EORTC HN35 questionnaires (patient reported outcome) will be evaluated
Identification of cytokine and growth factors | 36 months
  Identification of cytokines and growth factors in blood and their change during the course of dietary intervention; comparison with control arm; Identification of tumor DNA in saliva and blood
Monitoring of DNA methylation | 36 months
  The monitoring of DNA methylation obtained from salivary rinses in the 2 groups will help to identify biomarkers associated to the outcome of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Licitra, MD, Principal Investigator — Fondazione IRCCS Istituto Tumori Milano
Locations (6):
- Medical University of Vienna, Vienna, Austria
- Klinik und Poliklinik für Hals-, Nasen-, Ohrenheilkunde, Leipzig, Germany
- Fondazione IRCCS Istituto Nazionale Tumori, Milan, Lombardy, Italy
- The Greater Poland Cancer Centre, Poznan, Poland
- Grupo de Estudos de Cancro da Cabeça e Pescoço, Lisbon, Portugal
- Institute of Oncology Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No
The final results of the clinical study will be published in an impacted scientific journal.